CLINICAL TRIAL: NCT02155413
Title: Retrospective Study to Evaluate the Tolerability and Safety of Acute Pain Service at Queen Mary Hospital Between 2009 to 2012
Brief Title: Audit of Tolerability and Safety of Acute Pain Service
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cheung Chi Wai, Clinical Associate Professor, The University of Hong Kong
Other Study IDs: UW14-284
Record Dates: First submitted 2014-06-02; First posted 2014-06-04 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Acute Pain
Keywords: Acute pain; Audit; Safety; Tolerability
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Acute pain service (APS) was introduced in 1990s at Queen Mary Hospital (QMH) as other countries. With accumulation of experience and clinical evidence, APS has been well established. A study conducted in 1997 suggested that monitoring, management protocol and nursing experience were mandatory to the safety for APS. Our recent study showed that pain relief of our post-operative patients using patient controlled analgesic with morphine was still not adequate. The results has driven us to continue the improvement of post-operative outcomes for our surgical patients. Tolerability and safety are always our concerns for patients using our APS. Therefore, the investigators aim to conduct this retrospective study in order to assess if the tolerability and safety of our present APS are adequate or not. The study results will help us to further improve our APS at QMH if necessary.

DETAILED DESCRIPTION:
Retrospective audit.

Acute pain service records at Division of Pain Management, Department of Anaesthesiology, Queen Mary Hospital will be identified, validated and analysed.

Data Collection

1. Demographic data
2. Type of operation
3. Type of pain relief modality
4. Pain score up to 72 hours postoperatively
5. Types of operations and clinical variables
6. Incidence of adverse events during APS care;
7. Patients safety (ie respiratory depression)

Data Analysis For summarising analysis, mean or median with standard deviation or interquartile range will be reported. Parametric and non-parametric comparative tests will be used for analysis between/among patients with various characteristics. Kaplan Meier survival analysis and log-rank test will be used for duration of APS use.

ELIGIBILITY:
Inclusion Criteria:

* Postoperative patients who were cared by the Acute Pain Service, Pain Management Team, Department of Anaesthesiology, Queen Mary Hospital between 2009 to 2012.

Exclusion Criteria:

* Essential data were missing;
* Patient participating in other research projects.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Postoperative patients who were cared by the Acute Pain Service, Pain Management Team, Department of Anaesthesiology, Queen Mary Hospital between 2009 to 2012.
Sampling Method: Non-Probability Sample
Enrollment: 7500 (Estimated)
Dates: Start 2014-06; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Pain score | From postoperative 1 hour to postoperative 72 hour

SECONDARY OUTCOMES:
Incidence of adverse events | From postoperative 1 hour to postoperative 72 hour

OTHER OUTCOMES:
Incidence of serious adverse events (i.e respiratory depression) | From Post-operative day 1 to post-operative day 3

CONTACTS AND LOCATIONS:
Overall Officials: Chi Wai Cheung, MD, Principal Investigator — Department of Anaesthesiology, The University of Hong Kong
Locations (1):
- Department of Anaesthesiology, The University of Hong Kong, Hong Kong, Hong Kong